CLINICAL TRIAL: NCT03500588
Title: Vascular Endothelial Growth Factor C/A 2578 Gene Polymorphism and Umbilical Artery Doppler in Preeclamptic Women
Brief Title: Vascular Endothelial Factor Gene Polymorphism in Preeclampsia
Status: Completed | Type: Observational
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Nesreen Abdel Fattah Abdullah Shehata, Assistant professor, Beni-Suef University
Other Study IDs: BeniSuef 15
Record Dates: First submitted 2018-04-10; First posted 2018-04-18 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Ultrasonography, Doppler

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- normotensive pregnant women more than 20 weeks gestation.: One hundred and forty-five pregnant women after 20 weeks with normal blood pressure were evaluated for VEGF gene mutation.
  Interventions: Diagnostic Test: PCR
- Pregnant women after 20 weeks with preeclampsia.: One hundred and forty-five pregnant women after 20 weeks with preeclampsia were evaluated for VEGF gene mutation by using PCR and Pulsitality index of umbilical artery by doppler velocimetry.
  Interventions: Diagnostic Test: PCR; Device: Doppler ultrasound

INTERVENTIONS:
Diagnostic Test: PCR — Polymerase chain reaction was used to diagnose gene polymorphism.
Device: Doppler ultrasound — Doppler ultrasound was used to assess the pulsatility index of the umbilical artery .
  Groups: Pregnant women after 20 weeks with preeclampsia.

SUMMARY:
In this study, the investigators assessed one of the released protein factors during the pathophysiology of preeclampsia. They evaluated vascular endothelial growth factor gene mutation which affects the angiogenesis in case of inadequate placentation and its association with Doppler changes in the pulsatility index of the umbilical artery.

DETAILED DESCRIPTION:
Preeclampsia is a syndrome characterized by occurrence of hypertension and proteinuria after 20 weeks of gestation. The pathophysiology of preeclampsia involves abnormalities in the development of placental vasculature early in pregnancy may result in relative placental under perfusion/hypoxia/ischemia, which then leads to release of factors into the maternal circulation that alter maternal endothelial function and cause hypertension and other manifestations of disease .Vascular endothelial growth factor (VEGF) is a signal protein produced by cells that stimulates vasculogenesis and angiogenesis. It is part of the system that restores the oxygen supply to tissues when blood circulation is inadequate. Human VEGF gene is located on chromosome 6 and consists of 8 exons with alternate splicing, forming a family of proteins. There are several common single nucleotide polymorphisms (SNPs) in the VEGF gene, which could alter gene expression and protein production, and alter the risk of developing diseases characterized by deranged angiogenesis including preeclampsia.

ELIGIBILITY:
Inclusion Criteria:

More than 20 weeks gestation. Preeclamptic patients

Exclusion Criteria:

association with chronic disease (cardiac, hepatic, renal) and if the patient was known to have chronic hypertension.

association with auto-immune disease.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: normal and preeclamptic pregnant women after 20 weeks were evaluated for VEGF gene polymorphism.
Sampling Method: Probability Sample
Enrollment: 290 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Correlation of VEGF gene mutation and preeclampsia | from 20 weeks until delivery
  Is VEGF gene polymorphism associated with preeclampsia

SECONDARY OUTCOMES:
fetal and neonatal outcomes | from 20 weeks until first postpartum week.
  Intrauterine growth restriction
maternal outcome | from 20 weeks until delivery
  Maternal admission to intensive care unit

CONTACTS AND LOCATIONS:
Locations (1):
- Beni-Suef University, Cairo, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lain KY, Roberts JM. Contemporary concepts of the pathogenesis and management of preeclampsia. JAMA. 2002 Jun 26;287(24):3183-6. doi: 10.1001/jama.287.24.3183. No abstract available. PMID 12076198
- [Background] Huppertz B. Placental origins of preeclampsia: challenging the current hypothesis. Hypertension. 2008 Apr;51(4):970-5. doi: 10.1161/HYPERTENSIONAHA.107.107607. Epub 2008 Feb 7. No abstract available. PMID 18259009
- [Background] Cooper ME, Vranes D, Youssef S, Stacker SA, Cox AJ, Rizkalla B, Casley DJ, Bach LA, Kelly DJ, Gilbert RE. Increased renal expression of vascular endothelial growth factor (VEGF) and its receptor VEGFR-2 in experimental diabetes. Diabetes. 1999 Nov;48(11):2229-39. doi: 10.2337/diabetes.48.11.2229. PMID 10535459
- [Background] Chedraui P, Solis EJ, Bocci G, Gopal S, Russo E, Escobar GS, Hidalgo L, Perez-Lopez FR, Genazzani AR, Mannella P, Simoncini T. Feto-placental nitric oxide, asymmetric dimethylarginine and vascular endothelial growth factor (VEGF) levels and VEGF gene polymorphisms in severe preeclampsia. J Matern Fetal Neonatal Med. 2013 Feb;26(3):226-32. doi: 10.3109/14767058.2012.733760. Epub 2012 Oct 18. PMID 23039092